CLINICAL TRIAL: NCT06456801
Title: Clinical Trial of Anti-PLA2R-IgG Detection Kit (Time-resolved Fluorescence Immunoassay)
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Du Xiaoying, Department of nephrology, Zhejiang University
Other Study IDs: zjbs-pla2r-2012
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Nephropathy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Conduct comparative experimental studies on clinical serum samples using assessment reagents and approved products, and evaluate the equivalence between assessment reagents and comparison reagents.

DETAILED DESCRIPTION:
Conduct comparative experimental studies on clinical serum samples using assessment reagents and approved products, and evaluate the equivalence between assessment reagents and comparison reagents.

ELIGIBILITY:
Inclusion Criteria:

Clear background information and traceable sources of samples from kidney disease patients (number, age, gender, and clinical diagnostic information).

Exclusion Criteria:

Exclude serum samples that meet one of the following conditions:

① Samples with insufficient sample size, ② Samples with incomplete sample information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic kidney disease
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Calculate the correlation between the test reagents and comparison reagents | 1 year.
  Calculate the correlation between the test reagents and comparison reagents

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Du, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated hospital Zhejiang University school of medicine, Hangzhou, Zhejiang, China